CLINICAL TRIAL: NCT01847807
Title: The Cardiac and Kidney Protection of Astragalus in Subjects With Metabolic Syndrome
Brief Title: The Organ Protection of Astragalus in Subjects With Metabolic Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LanZhou University (Other)
Responsible Party: Principal Investigator, Jing Yu, cheif of cardiology, LanZhou University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS2304
Record Dates: First submitted 2013-05-02; First posted 2013-05-07 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Metabolic Syndrome
Keywords: 5-10 gram astragalus per day
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High-dose Astragalus group (Active Comparator): treatment with 10 gram astragalus
  Interventions: Drug: high dose astagalus
- Low-dose Astragalus group (Active Comparator): treatment with 5 gram astragalus
  Interventions: Drug: low dose Astragalus
- MS control (No Intervention)

INTERVENTIONS:
Drug: low dose Astragalus
  Arms: Low-dose Astragalus group
Drug: high dose astagalus
  Arms: High-dose Astragalus group

SUMMARY:
Metabolic syndrome have the damages on tissues and organs in heart、kindey and vessels. In this study, prospective randomized, controlled, parallel designed ,different doses of Astragalus Mongolia, Gansu Longxi produce treat on the MS patients, and then use real-time quantitative PCR and Western Blotting to detect the index of oxidative stress 、angiotensin-converting enzyme 2 mRNA expression and proteins.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 years or older, meet the diagnostic criteria of MS
2. non-allergic with the astragalus
3. agree to conduct clinical trials and those who signed the informed consent

Exclusion Criteria:

1. patients with resistant hypertension
2. renal disease requiring dialysis
3. heart failure NYHA ⅢorⅣ;
4. complications of diabetes
5. arteritis
6. cancer
7. thyroid disease
8. unstable coronary heart disease
9. peripheral vascular disease
10. acute cerebral vascular disease11.pregnancy、 planned pregnancy
11. patients with anti-oxidants
12. acute infection
13. other organic dysfunction, such as the liver, respiratory system, blood system, and other rheumatic diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2011-01; Primary Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
index of cardiac function | one year
  ues echocardiography to measure the cardiac function

SECONDARY OUTCOMES:
blood pressure | one year

OTHER OUTCOMES:
kidney function | one year
Central Blood Pressure | one year
Ankle Brachial Index | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Lanzhou University Second Hospital, Lanzhou, Gansu, China